CLINICAL TRIAL: NCT02097199
Title: Influence of Physical Activity on Promising Atherosclerosis Biomarkers
Brief Title: IPHAAB-study Influence of Physical Activity on Atherosclerosis Biomarkers
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Collaborators: Austrian Federal Ministry of Defence and Sports (Unknown)
Responsible Party: Principal Investigator, Jeanette Strametz-Juranek, Prim.Univ.Prof.Dr., Medical University of Vienna
Other Study IDs: 1830/2013
Record Dates: First submitted 2014-03-24; First posted 2014-03-26 (Estimated); Last update posted 2016-01-07 (Estimated); Status verified 2016-01

CONDITIONS: Influence of 8 Months of Increased Physical Activity Workload on Osteoprotegerin and Endocan Levels
Keywords: activity, osteoprotegerin, endocan, atherosclerosis, biomarker
MeSH Terms: conditions — Motor Activity; Atherosclerosis

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — whole blood
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Sports group: The cohort will consist of about 55 female and 55 male individuals aged 30-65 years with mostly sedentary work (>6 hours/day) doing no or less physical activity (<30 minutes quick walking/day) who want to engage more in physical activity (at least 150 minutes of at least moderate intensity per week). The gain in workload will be objectified and quantified by performing a bicycle stress test at the beginning of the study and after 8 months of physical engagement.
  Interventions: Other: Increased sports workload

INTERVENTIONS:
Other: Increased sports workload — At least 150 minutes of moderate or 75 minutes of vigorous exercise per week. The "Recommendations for Adults From the American College of Sports Medicine and the American Heart Association" clearly define physical exercise intensity levels. The present study follows these recommendations. Consequently, moderate physical activity can be reached by e.g. quick walking, slow bicycling, slow swimming...; it is also possible to reach the expected workload by engaging in vigorous exercise (e.g. jogging/running, quick swimming, playing soccer/tennis...). The gain in performance will objectified by performing a bicycle stress test at the beginning and the end of the study.

SUMMARY:
This study investigates the influence of an increased physical activity and sports workload in formerly nonsporting healthy individuals on current promising biomarkers of atherosclerosis research.

DETAILED DESCRIPTION:
According to Statistik Austria, cardiovascular disease (CVD) is the most common reason for death in Austria in total population. In 2011, 42,3 % of all deaths were due to CVD (ICD-10 I00-I99). In People aged 45-64 years, CVD is, beyond cancer, the second most common cause of death. According to the "Österreichische Gesundheitsbefragung 2006/7" more than two-thirds of men and three-quarters of women are physically inactive whereby physical inactivity was defined as at least 3x/week of sudatory exercise like cycling, jogging or aerobic.

A very famous study done by Morris et al. in 1953 showed that bus conductors in London (walking job) had half of the coronary heart disease (CHD) mortality compared to bus drivers (sitting job) and therefore initiated the hour of birth of CVD research in connection to physical (in)activity. Cardiorespiratory fitness might reduce does-dependently all cause cardiovascular mortality by 20-30 % (5-8) and the probability of developing CHD by 30-50 % (9-11).

Recently, CVD-research focuses on the investigation of blood-markers which indicate the presence of atherosclerosis and represent risk for development and genesis of CV events. E.g. inflammatory markers such as IL-6, TNF-alpha, ICAM-1, P-selectin, hsCRP and serum amyloid A are promising markers. Studies have shown that hsCRP levels at baseline predict future CV events. Markers of plaque stability are e.g. myeloperoxidase, metalloproteinase-9 and soluble CD-40 ligand. However, the influence of exercise on these factors has already been investigated.

The main dependent variables will be endocan and osteoprotegerin (OPG): OPG is a member of the TNF-related family and involved in bone metabolism. However, high levels of OPG have been reported in association with cardiovascular outcome (CAD, vascular calcification, advanced atherosclerosis, heart failure...). Serum concentrations were found to correlate with severity of peripheral artery disease, carotic stenosis and myocardial infarction. Furthermore, OPG is was associated with left ventricle and left atrial remodelling in patients with severe aortic stenosis, a disease which is often obverse in elderly patients. Age and gender were shown to predict OPG levels, at least in hemodialysis patients. Several studies have been performed investigating the influence of acute exercise or resistance training on circulating OPG amounts but less is known about the influence of long-term physical exercise.

Endocan (endothelial cell specific molecule 1; ESM-1) is a recombinant proteoglycan which may represent a new marker that correlates with CV risk and surrogate endothelial dysfunction playing a role in endothelium-dependent pathological disorders.

Other variables will be:

* Progerin: Progerin was originally investigated in course of research in Hutchinson-Gilford-Syndrome, a genetic effect which affects children leading to atherosclerosis. Progerin correlates with the vascular pathology of "normal" aging and is present also in the "normal" population.
* Myeloid-related protein 8 and 14 (MRP-8/14): MRP-8/14 is a stable heterodimer, formed by Ca++-binding proteins. It has been shown that MRP-8/14 regulates vascular inflammation, is involved in diabetic vascular complications and occurs in CAD. Furthermore, MRP-14 was associated with histopathologic findings and inflammation status in atherosclerotic plaques.
* Angiopoietin-like protein 2 (angptl2): Angptl2 depends to the family of angiopoietin-like proteins and is involved in angiogenesis. Angptl2 was shown to be 6 times higher in mice with CAD compared to controls. Furthermore, it increases with age but this increase was more pronounced in mice with high cholesterol levels. Angptl2 therefore contributes to the genesis and pathogenesis of atherosclerosis.
* Cathepsin S and K: Cathepsins are synthesized as inactive proenzymes and get activated by proteolytic processes. Atherosclerotic lesions contain much higher amounts of cathepsin S and K than normal arteries. Furthermore, they seem to play a role in the formation of aneurysms.
* Cystatin C: Cystatin C is a cysteine protease inhibitor participating in protein catabolism and has been suggested to predict CVD. High serum levels of cystatin c were shown to correlate with early stage atherosclerosis. Cystatin C is an independent predictor for the risk of cardiovascular events.
* Placental growth factor (PlGF): PlGF, a cysteine-knot protein which is quite homologous to VEGF, was implicated in the Pathophysiology of angiogenesis. PlGF-expression in atherosclerotic lesions was shown to be associated with inflammation and microvascular density suggesting PlGF to play a role in plaque destabilization and clinical manifestation of CAD (32). Anti-PlGF monoclonal antibody therapy in mice lead to a decrease in development of atherosclerosis.

All mentioned markers are of distinctive interest in atherosclerosis research, however, the influence of long-term exercise on them has not been studied yet.

ELIGIBILITY:
Inclusion Criteria:

* Age 30-65 years
* less than 30 minutes of quick walking/day
* Physical ability to perform sports and bicycle stress tests

Exclusion Criteria:

* Age <30 or >65 years
* Pregnancy
* weight >130 kg
* untreated/uncontrolled hypertension

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will consist of about 55 female and 55 male individuals aged 30-65 years with mostly sedentary work (>6 hours/day) doing no or less physical activity (<30 minutes quick walking/day).
Sampling Method: Non-Probability Sample
Enrollment: 98 (Actual)
Dates: Start 2014-08; Primary Completion 2015-11 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline osteoprotegerin and endocan level to osteoprotegerin and endocan levels after 8 months of increased physical activity workload | Baseline, Month 8
  Osteoprotegerin and endocan levels will be measured at baseline, every 2 months of training and at the end of the observation after 8 months

SECONDARY OUTCOMES:
Change from baseline Progerin, Myeloid-related peptide 8 and 14, Angiopoietin-like protein 2, Cathepsin S and K, Cystatin C and Placental growth factor level to levels after 8 months of increased physical activity workload | Baseline, Month 8
  Progerin, Myeloid-related peptide 8 and 14, Angiopoietin-like protein 2, Cathepsin S and K, Cystatin C and Placental growth levels will be measured at baseline, every 2 months of training and at the end of the observation after 8 months

CONTACTS AND LOCATIONS:
Overall Officials: Jeanette Strametz-Juranek, Prof.Dr., Study Chair — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Vienna, Austria

REFERENCES:
- [Background] Sponder M, Dangl D, Kampf S, Fritzer-Szekeres M, Strametz-Juranek J. Exercise increases serum endostatin levels in female and male patients with diabetes and controls. Cardiovasc Diabetol. 2014 Jan 6;13:6. doi: 10.1186/1475-2840-13-6. PMID 24393402
- [Background] Sponder M, Sepiol K, Lankisch S, Priglinger M, Kampf S, Litschauer B, Fritzer-Szekeres M, Strametz-Juranek J. Endostatin and physical exercise in young female and male athletes and controls. Int J Sports Med. 2014 Dec;35(13):1138-42. doi: 10.1055/s-0034-1375692. Epub 2014 Jul 10. PMID 25009962
- [Background] Sponder M, Fritzer-Szekeres M, Marculescu R, Litschauer B, Strametz-Juranek J. Physical inactivity increases endostatin and osteopontin in patients with coronary artery disease. Heart Vessels. 2016 Oct;31(10):1603-8. doi: 10.1007/s00380-015-0778-6. Epub 2015 Dec 11. PMID 26661073
- [Derived] Lenz M, Schonbauer R, Stojkovic S, Lee J, Gatterer C, Lichtenauer M, Paar V, Emich M, Fritzer-Szekeres M, Strametz-Juranek J, Graf S, Sponder M. RANTES and CD40L under Conditions of Long-Term Physical Exercise: A Potential Link to Adaptive Immunity. Int J Environ Res Public Health. 2022 Jul 16;19(14):8658. doi: 10.3390/ijerph19148658. PMID 35886510
- [Derived] Sponder M, Lichtenauer M, Wernly B, Paar V, Hoppe U, Emich M, Fritzer-Szekeres M, Litschauer B, Strametz-Juranek J. Serum heart-type fatty acid-binding protein decreases and soluble isoform of suppression of tumorigenicity 2 increases significantly by long-term physical activity. J Investig Med. 2019 Jun;67(5):833-840. doi: 10.1136/jim-2018-000913. Epub 2018 Dec 27. PMID 30593542
- [Derived] Sponder M, Campean IA, Emich M, Fritzer-Szekeres M, Litschauer B, Graf S, Dalos D, Strametz-Juranek J. Long-term physical activity leads to a significant increase in serum sRAGE levels: a sign of decreased AGE-mediated inflammation due to physical activity? Heart Vessels. 2018 Aug;33(8):893-900. doi: 10.1007/s00380-018-1125-5. Epub 2018 Jan 24. PMID 29368166
- [Derived] Sponder M, Minichsdorfer C, Campean IA, Emich M, Fritzer-Szekeres M, Litschauer B, Strametz-Juranek J. Long-term endurance training increases serum cathepsin S levels in healthy female subjects. Ir J Med Sci. 2018 Aug;187(3):845-851. doi: 10.1007/s11845-017-1693-x. Epub 2017 Nov 27. PMID 29181829
- [Derived] Sponder M, Campean IA, Emich M, Fritzer-Szekeres M, Litschauer B, Bergler-Klein J, Graf S, Strametz-Juranek J. Endurance training significantly increases serum endocan but not osteoprotegerin levels: a prospective observational study. BMC Cardiovasc Disord. 2017 Jan 5;17(1):13. doi: 10.1186/s12872-016-0452-7. PMID 28056805